CLINICAL TRIAL: NCT01589458
Title: Fluoride Availability in Saliva After Use of NaF or MFP Toothpastes
Brief Title: Fluoride Availability in Saliva After Use of Sodium Fluoride or Monofluorophosphate Toothpastes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Livia Maria Andaló Tenuta, Assistant Professor, Biochemistry and Cariology, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FOPBioq003
Record Dates: First submitted 2012-04-29; First posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Dental Caries
Keywords: toothpastes; saliva; dental caries; fluoride
MeSH Terms: conditions — Dental Caries | interventions — Toothpastes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non-fluoride toothpaste (Placebo Comparator)
  Interventions: Drug: Toothpaste
- NaF/SiO2 toothpaste (Experimental)
  Interventions: Drug: Toothpaste
- MFP/CaCO3 toothpaste (Experimental)
  Interventions: Drug: Toothpaste

INTERVENTIONS:
Drug: Toothpaste — 1-min brushing with 1 g of the assigned toothpaste followed by a 10 mL purified water rinse

SUMMARY:
Considering the widespread use of sodium fluoride (NaF) and monofluorophosphate (MFP) based toothpastes, the present study aim to evaluate F availability in saliva after use of the top-selling Brazilian toothpastes. In a blind, crossover clinical trial study, volunteers will brush their teeth with one of the following toothpastes: 1) non-fluoride toothpaste (negative control group); 2) NaF/silica based toothpaste 3)MFP/calcium carbonate based toothpaste. After brushing, a rinse with purified water will be performed. Unstimulated saliva will be collected before and up to 60 min after brushing. Ionic fluoride and total soluble fluoride (corresponding to the sum of fluoride as ion and as MFP) will be determined after acid treatment of salivary samples to hydrolyze MFP. Fluoride will be determined using an ion selective electrode.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Good oral health
* Normal salivary flow rate

Exclusion Criteria:

* Use of systemic drugs that reduce salivary flow rate

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Area under the curve of salivary fluoride concentration versus time after brushing with fluoride toothpastes | 60 minutes

SECONDARY OUTCOMES:
Percentage of MFP hydrolyzed in saliva as a function of time | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Livia MA Tenuta, PhD, Principal Investigator — Piracicaba Dental School, University of Campinas
Locations (1):
- Piracicaba Dental School, University of Campinas, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Background] Cury JA, Tenuta LM, Ribeiro CC, Paes Leme AF. The importance of fluoride dentifrices to the current dental caries prevalence in Brazil. Braz Dent J. 2004;15(3):167-74. doi: 10.1590/s0103-64402004000300001. Epub 2005 Mar 18. PMID 15798817
- [Background] Ricomini Filho AP, Tenuta LM, Fernandes FS, Calvo AF, Kusano SC, Cury JA. Fluoride concentration in the top-selling Brazilian toothpastes purchased at different regions. Braz Dent J. 2012;23(1):45-8. doi: 10.1590/s0103-64402012000100008. PMID 22460314
- [Background] Cury JA, Oliveira MJ, Martins CC, Tenuta LM, Paiva SM. Available fluoride in toothpastes used by Brazilian children. Braz Dent J. 2010;21(5):396-400. doi: 10.1590/s0103-64402010000500003. PMID 21180793
- [Background] Tenuta LM, Cury JA. Fluoride: its role in dentistry. Braz Oral Res. 2010;24 Suppl 1:9-17. doi: 10.1590/s1806-83242010000500003. PMID 20857070
- [Background] Carrera CA, Giacaman RA, Munoz-Sandoval C, Cury JA. Total and soluble fluoride content in commercial dentifrices in Chile. Acta Odontol Scand. 2012 Dec;70(6):583-8. doi: 10.3109/00016357.2011.640287. Epub 2011 Dec 20. PMID 22182293